CLINICAL TRIAL: NCT00902499
Title: Evolution of Memory-related fMRI Activation Over the Course of MCI and AD
Brief Title: Evolution of Memory Related Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Reisa A. Sperling, MD, Brigham and Women's Hospital
Other Study IDs: IA0159; 5R01AG027435-04 (NIH)
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: functional magnetic resonance imaging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- NC: Normal older controls, not cognitively impaired; MMSE 27-30 and performance above education adjusted cutoff scores on the Logical Memory II subscale (LM-II Delayed Paragraph Recall) of the Wechsler Memory Scale
- vMCI: Very mild cognitive impairment; less severe objective memory deficit, scoring .5 to 1.5 S.D. (standard deviation) below education adjusted norms on the LM-II
- sMCI: significant mild cognitive impairment; objective cut off of 1.5 S.D. level below education adjusted norms on the LM-II
- AD: Mild Alzheimer's disease; meet NINCDS/ADRDA criteria for probable AD with mild dementia severity (CDR Total = 1), MMSE 20-26

SUMMARY:
The purpose of this study is to begin the process of validating fMRI (functional magnetic resonance imaging) as a biomarker for use in clinical trials and longitudinal studies of clinical progression in mild cognitive impairment (MCI) and Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The development of biomarkers is now especially critical, as there are a number of promising disease-modifying therapies entering early phase clinical trials, with additional novel therapeutic strategies in development. It is essential to develop biomarkers that can detect a "signal of efficacy" over a relatively short time frame for use in Phase II trials. Ideally biomarkers are needed that can reliably detect the earliest brain alterations due to AD pathology, perhaps at a point when there is synaptic dysfunction but not yet widespread neuronal loss. Functional neuroimaging, in particular functional MRI (fMRI), has significant potential, having already shown promise in detecting regionally specific pharmacological effects on memory related neural activity, and as a sensitive marker of very early cognitive impairment.

This study, a parallel ancillary study of the Alzheimer's Disease Neuroimaging Initiative (ADNI), will first examine reproducibility of fMRI activation, using a face-name associative memory paradigm, and then the alterations in memory-related activation that occur over the course of MCI and mild AD. The study will also examine the relationship of fMRI activation to clinical variables, memory task performance, genotype, and other imaging techniques cross-sectionally and longitudinally, sampling at multiple time points over a 3-year period.

ELIGIBILITY:
Inclusion Criteria:

* Ages 55-90
* General good health or stable medical problems
* Study partner/caregiver able to provide an independent evaluation of the participant's daily functioning
* No contraindications to MR scanning
* Modified Hachinski Ischemic Score ≤4
* Geriatric Depression Scale ≤10

Exclusion Criteria:

* Diagnosis of Parkinson's disease or other neurological illness
* Presence of clinically significant/uncontrolled medical conditions
* History of stroke, brain tumor, brain surgery, seizures, significant head trauma with loss of consciousness, depression or other psychiatric illness, alcohol or drug abuse in the past 2 years
* Significant uncorrectable visual impairment

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Memory Disorders Unit at Brigham and Women's Hospital, the Gerontology Research Unit at Massachusetts General Hospital, Alzheimer's Association, area physicians, and community dwelling adults
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2006-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Reisa Sperling, MD, Principal Investigator — Director of Clinical Research, Memory Disorders Unit, Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Sperling R, Greve D, Dale A, Killiany R, Holmes J, Rosas HD, Cocchiarella A, Firth P, Rosen B, Lake S, Lange N, Routledge C, Albert M. Functional MRI detection of pharmacologically induced memory impairment. Proc Natl Acad Sci U S A. 2002 Jan 8;99(1):455-60. doi: 10.1073/pnas.012467899. Epub 2001 Dec 26. PMID 11756667
- [Background] Sperling RA, Bates JF, Chua EF, Cocchiarella AJ, Rentz DM, Rosen BR, Schacter DL, Albert MS. fMRI studies of associative encoding in young and elderly controls and mild Alzheimer's disease. J Neurol Neurosurg Psychiatry. 2003 Jan;74(1):44-50. doi: 10.1136/jnnp.74.1.44. PMID 12486265
- [Background] Greicius MD, Srivastava G, Reiss AL, Menon V. Default-mode network activity distinguishes Alzheimer's disease from healthy aging: evidence from functional MRI. Proc Natl Acad Sci U S A. 2004 Mar 30;101(13):4637-42. doi: 10.1073/pnas.0308627101. Epub 2004 Mar 15. PMID 15070770
- [Background] Grundman M, Petersen RC, Ferris SH, Thomas RG, Aisen PS, Bennett DA, Foster NL, Jack CR Jr, Galasko DR, Doody R, Kaye J, Sano M, Mohs R, Gauthier S, Kim HT, Jin S, Schultz AN, Schafer K, Mulnard R, van Dyck CH, Mintzer J, Zamrini EY, Cahn-Weiner D, Thal LJ; Alzheimer's Disease Cooperative Study. Mild cognitive impairment can be distinguished from Alzheimer disease and normal aging for clinical trials. Arch Neurol. 2004 Jan;61(1):59-66. doi: 10.1001/archneur.61.1.59. PMID 14732621